CLINICAL TRIAL: NCT00002632
Title: PHASE II TRIAL OF TAXOL IN ADVANCED OR METASTATIC SALIVARY GLAND MALIGNANCIES
Brief Title: Paclitaxel in Treating Patients With Metastatic or Recurrent Salivary Gland Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064057; E-1394
Record Dates: First submitted 1999-11-01; First posted 2004-06-10 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Cancer
Keywords: stage IV salivary gland cancer; recurrent salivary gland cancer; high-grade salivary gland mucoepidermoid carcinoma; salivary gland adenocarcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of paclitaxel in treating patients with metastatic or recurrent salivary gland cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the response rate in patients with metastatic or recurrent salivary gland cancer treated with paclitaxel (Taxol, TAX) by 3-hour infusion. II. Describe the toxicity of TAX in these patients.

OUTLINE: Single-Agent Chemotherapy. Paclitaxel (Bristol-Myers), Taxol, TAX, NSC-125973.

PROJECTED ACCRUAL: Up to 32 patients/histology will be entered. If no response is observed in the first 14 patients in a particular histology, accrual to that group will close; if after 18 months annual accrual is less than 10 patients/histology, accrual to that group may close.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed salivary gland carcinoma that is metastatic or recurrent, including the following types: Mucoepidermoid carcinoma Adenocarcinoma Pathology review required Measurable disease required Lesion in a previously irradiated field must be progressing and biopsy- proven

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Hematopoietic: WBC at least 3,000/mm3 ANC at least 1,500/mm3 Platelet count at least 100,000/mm3 Hb at least 10 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No MI within the past 6 months No CHF No unstable arrhythmia No current antiarrhythmic, inotropic, or antianginal medication Other: No history of allergy to Cremophor No prior malignancy within 5 years except: Curatively treated nonmelanomatous skin cancer Curatively treated in-situ cancer of the cervix No concurrent malignancy Not pregnant or nursing Effective contraception strongly advised for fertile patients Blood/body fluid analyses to determine eligibility and imaging studies and scans/x-rays for tumor measurement completed within 14 days prior to registration

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior biological response modifier therapy allowed Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed with recovery Surgery: Prior surgery allowed with recovery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 1995-05-30 (Actual); Primary Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harlan A. Pinto, MD, Study Chair — Stanford University
Locations (29):
- United States (28):
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Lakeside), Chicago, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Nashville, Nashville, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Gilbert J, Li Y, Pinto HA, Jennings T, Kies MS, Silverman P, Forastiere AA. Phase II trial of taxol in salivary gland malignancies (E1394): a trial of the Eastern Cooperative Oncology Group. Head Neck. 2006 Mar;28(3):197-204. doi: 10.1002/hed.20327. PMID 16470745
- [Result] Jennings T, Li Y, Pinto H, et al.: Phase II trial of paclitaxel in advanced or metastatic salivary gland malignancies: an Eastern Cooperative Oncology Group study. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-942, 2001.